CLINICAL TRIAL: NCT05890781
Title: Engineering Immune Organoids to Study Pediatric Cancer (IMMUNE-ORGANOIDS)
Brief Title: Engineering Immune Organoids to Study Pediatric Cancer
Acronym: IMMUNEORGANOID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A03021-38; 2020/3712 (Other: CSET number)
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brain Tumor; Kidney Tumor; Neuroblastoma; Sarcoma
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Renal Cell; Neuroblastoma; Sarcoma | interventions — Blood Specimen Collection; Cerebrospinal Fluid Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immune organoids from pediatric patient tissues using iPSC (Other): To engineer immune organoids from pediatric patient tissues using induced-pluripotent stem cells (iPSC)
  Interventions: Procedure: Skin biopsy; Procedure: Fresh tumor sample; Biological: Blood sample; Procedure: Healthy tissue from the tumor; Procedure: Spinal cerebrospinal fluid (SCF)

INTERVENTIONS:
Procedure: Skin biopsy — Skin biopsy
Procedure: Fresh tumor sample — Fresh tumor sample
Biological: Blood sample — Blood sample in heparin tubes (highly recommended), to be collected before starting treatment or as soon as hematological recovery has been reached
Procedure: Healthy tissue from the tumor — Healthy tissue from the tumor site whenever possible
Procedure: Spinal cerebrospinal fluid (SCF) — Spinal cerebrospinal fluid (SCF) whenever possible

SUMMARY:
To engineer immune organoids from pediatric patient tissues using induced-pluripotent stem cells (iPSC)

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis ≤ 25 years except for patients with malignant gliomas and renal tumors for whom no upper age limit is applied
* Medical suspicion or diagnosis of one of the following diseases, regardless of stage:
* Brain tumors
* Renal tumors
* Neuroblastoma
* Sarcomas
* Adult patient or parents or guardians should understand, sign and date the appropriate written informed consent from prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

* Any histology not mentioned in the inclusion criteria
* Adult patient or parents/guardians incapable/incapable of giving its/their consent
* Patients deprived of their liberty by a judicial or administrative decision

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of viable and exploitable immune organoids with engrafted tumor cells | until 5 years after enrolment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Gustave Roussy, Villejuif
  - Hopital Necker, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided